CLINICAL TRIAL: NCT03192293
Title: Single Arm Phase 2 Study of Metformin and Simvastatin in Addition to Fulvestrant in Metastatic Estrogen Receptor Positive Breast Cancer
Brief Title: Metformin and Simvastatin in Addition to Fulvestrant
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BR03/10/16; 2016/01178 (Other: NHG DSRB)
Record Dates: First submitted 2017-02-06; First posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metformin/Simvastatin/Fulvestrant (Experimental): 7 days Lead-in period:
  1. Metformin: 850mg (one tablet) twice a day
  2. Simvastatin: 20mg (one tablet) once every night
  Once the doctor has deemed that patients have tolerated Simvastatin and Metformin well, patients will receive Fulvestrant at standard doses:
  1. Cycle 1: 500mg (in the form of two injections, 1 in each buttock) at Day 1 and Day 15. Each cycle comprises of 28 consecutive days starting from Day 1.
  2. Cycle 2 and beyond: 500mg at Day 1 of each 28-day cycle.
  Interventions: Drug: Metformin/Simvastatin/Fulvestrant

INTERVENTIONS:
Drug: Metformin/Simvastatin/Fulvestrant — 7 days Lead-in period: Metformin: 850mg (one tablet) twice a day Simvastatin: 20mg (one tablet) once every night
  Once the doctor has deemed that patients have tolerated Simvastatin and Metformin well, patients will receive Fulvestrant at standard doses:
  Cycle 1: 500mg (in the form of two injections, 1 in each buttock) at Day 1 and Day 15. Each cycle comprises of 28 consecutive days starting from Day 1.
  Cycle 2 and beyond: 500mg at Day 1 of each 28-day cycle.
  Tumour biopsy at 8 weeks. Every 8 weeks for the first 6 months, every 12 weeks thereafter:
  Performance status evaluation Medical history and physical examination Clinical tumor measurement Review of treatment-related side-effects Blood taking for research purpose and routine blood tests Routine scans

SUMMARY:
This is a prospective single arm open-label Phase 2 study utilising the combination of Fulvestrant, Metformin and Simvastatin in post-menopausal ER-positive metastatic breast cancer, with the primary endpoint being Clinical Benefit Rate (defined as complete response, partial response or stable disease, equal to or more than 24 weeks). The hypothesis is that the addition of Metformin and Simvastatin to Fulvestrant will improve the Clinical Benefit Rate from 40% (historical data from control arm of PALOMA-3 study) to 60%. A total of 28 patients will be enrolled over a period of 24 months. Eligible patients will receive 500 mg Fulvestrant by intramuscular injection on days 1 and 15 of cycle one and then on day one of each subsequent cycle (28 days). Patients will be given 850mg oral Metformin twice-a-day (based on xenograft models which showed that Metformin had anti-tumor effects at a minimum dose of 1500mg per day), and 20mg oral Simvastatin every night (drawing reference from the investigators' group's window-of-opportunity study), daily throughout the cycle. As part of the in-build safety and tolerability design, all patients will have a lead-in period of 7 days where they receive 850mg oral Metformin twice-a-day and 20mg oral Simvastatin every night. Special adverse events of interest include lactic acidosis, diarrhea, bloatedness, transaminitis and rhabdomyolysis. If no dose-limiting toxic effects (DLT) occur, Fulvestrant will be commenced, and considered the start of cycle 1. If DLT occurs in any of the patients, the combination of Metformin and Simvastatin will be modified for the affected patient as per protocol, with further monitoring for another 7 days. This combination will be deemed safe for that patient if no DLT occurs, following which cycle 1 can officially commence.

At the time of study entry, blood samples will be drawn to establish baseline physiological parameters including fasting insulin, glucose, lipids and Homeostasis Model Assessment 2 (HOMA2). In patients who have accessible tumor sites and are willing to provide tissue for translational research, pre- and post-treatment (at end of 8 weeks) biopsies will be taken for correlative biomarker studies. Patients will be evaluated on an 8-weekly basis for toxicities and efficacy assessments during the first 6 months of treatment, followed by 12-weekly thereafter until disease progression, unacceptable toxicities, or patient withdrawal.

DETAILED DESCRIPTION:
Endocrine therapy and acquired endocrine resistance in advanced breast cancer:

First-line treatment of metastatic estrogen receptor (ER) positive breast cancer with endocrine therapy such as Tamoxifen or aromatase inhibitors (AI) is efficacious, but development of secondary resistance is inevitable with median progression free survival of 9 months.1 Acquired resistance can be contributed by molecular cross-talk between estrogen receptors and other key survival and proliferative pathways. In particular, the PI3K/Akt/MAP kinase signaling pathway is upregulated with prolonged estrogen deprivation and is an important feature of progressive disease biology.2

The BOLERO-2 study showed an improvement in response rates and progression free survival with the addition of Everolimus, an mTOR-inhibitor to Exemestane in metastatic ER-positive breast cancer after failure on a non-steroidal AI.3 Synergy was also seen in a Phase 2 clinical trial with the combination of Fulvestrant and Everolimus in the second line setting.4 However, the clinical experience with Everolimus has been poor, with frequent adverse effects rendering the combination with endocrine therapy highly toxic. More recently, the PALOMA-1/3 studies have showed that targeting the CDK4/CDK6/E2F axis with Palbociclib is a feasible strategy with marked improvements in clinical endpoints when combined with Letrozole in the first line, and Fulvestrant after AI-failure.5,6 While the therapy was reasonably well-tolerated, Palbociclib remains prohibitively expensive, and is not widely used in countries where healthcare systems do not cover the cost of this novel combination.

Potential of Metformin and Simvastatin as anti-cancer agents:

It has been widely recognized that Metformin and Simvastatin, both commonly used medications in diabetes mellitus and dyslipidemia, have anti-cancer properties. Years of experience in the real world have shown that at standard doses, these 2 drugs can be used in combination with little toxicities. Metformin, a biguanide, results in activation of AMPK which consequently inhibits mTOR through phosphorylation of TSC2, as well as anti-proliferative effects through reduction in insulin receptor mediated mitogenesis and inhibition of cyclin dependent kinases.7,8 Pre-clinical studies in mouse xenograft models showed that at an equivalent dose of at least 1500mg per day, Metformin reduced the effective dosage of standard chemotherapeutic agents, and had preferential effects on tumor cells.9 Studies of Metformin in MCF7, an ER-positive breast cancer cell line, also showed that it resulted in significant reduction in protein synthesis as well as inhibition of the mTOR pathway.10 Simvastatin, a lipophilic HMGCoA reductase inhibitor, has been shown to interrupt oncogenic signaling by prenylation-dependent proteins including the RAS oncogene family, and attenuate PI3K signaling. In a recent window-of-opportunity study by the inverstigators' group, the investigators showed that at the usual prescribed dose of Simvastatin (20mg), a short course of therapy resulted in evident apoptosis and de-activation of the PI3K/Akt/mTOR and MAPK/ERK pathways in both clinical specimens as well as breast cancer cell lines.12

The investigators believe that there is untapped potential in the usage of Metformin and Simvastatin in targeting the PI3K/Akt/mTOR pathway which is upregulated in metastatic ER-positive breast cancer after progression on first-line endocrine therapy, and that this inexpensive and non-toxic combination will show synergy with Fulvestrant in the second-line (and beyond) setting.

ELIGIBILITY:
Eligibility criteria:

* Women 18 years or older with metastatic or locally advanced disease, not amenable to curative therapy
* Confirmed diagnosis of HR+/HER2- breast cancer
* Any menopausal status
* Progressed within 12 months from prior adjuvant or progressed within 1 month from prior advanced/metastatic endocrine breast cancer therapy
* On an LHRH agonist for at least 28 days, if pre-/peri-menopausal*.
* Measurable disease defined by RECIST version 1.1, or bone-only disease
* Eastern Cooperative Oncology Group (ECOG) PS 0-2 and estimated life expectancy of at least 12 weeks
* Adequate organ and marrow function, resolution of all toxic effects of prior therapy or surgical procedures
* Signed informed consent
* Pre-menopausal* females must have a negative serum pregnancy test within 21 days of study enrollment

  * Definition of Menopause:

    i. Age > 60 years, ii. Age < 60 years with amenorrhoea for > 12 months in the absence of endocrine therapy or chemotherapy iii. Bilateral oophorectomy

Exclusion criteria:

* Prior treatment with any CDK inhibitor, Fulvestrant, Everolimus, or agent that inhibits the PI3K-mTOR pathway
* Patients with symptomatic visceral disease, or known uncontrolled or symptomatic CNS metastases
* Patients who have not yet recovered from the toxicities of the previous anti-cancer therapy.
* Concurrent administration of other anti-tumor therapies, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy are prohibited. Concomitant bone-modifying agents and gonadotropin-releasing hormone therapy are allowed.
* Major surgery or radiotherapy within 2 weeks of randomization
* Prior stem cell or bone marrow transplantation
* Use of potent CYP3A4 inhibitors or inducers (Table 1); a washout period of 14 days is required for patients discontinuing these medications prior to study enrollment.
* Currently on medications for diabetes (e.g. Metformin, sulphonylureas, insulin) or hypercholesterolaemia (statins or fibrates)
* Renal impairment: Estimated glomerular filtration rate (eGFR) <60 mL/minute/1.73 m2
* Hepatic impairment: Aspartate transaminase (AST), Alanine Transaminase(ALT) ≥ 2.5 x upper limit of normal range (ULN), OR Total bilirubin ≥ 1.5 x ULN (subjects with Gilbert's syndrome can have bilirubin of up to 1.5 x ULN)
* Pregnancy.
* Breast feeding.
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 28 (Estimated)
Dates: Start 2017-01-20 (Actual); Primary Completion 2019-01-20 (Estimated); Study Completion 2019-01-20 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit rate (CBR) | The Clinical Benefit Rate will be assessed at 24 weeks of treatment with study drug. The time frame will be through study completion, in an average of 2 years.
  the percentage achieving CR, PR and SD in patients with measurable disease or the absence of disease progression in patients with non-measurable disease, lasting at least 24 weeks.

SECONDARY OUTCOMES:
Objective response rates (ORR) | The Objective Response Rate will be assessed from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed through study completion, in an average of 2 years.
  a best overall response of CR or PR.
Progression-free survival (PFS) | The progression-free survival will be assessed from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed through study completion, in an average of 2 years.
  the time from the date of study enrollment until the first date of documented disease progression or death due to any cause, whichever occurs first.
Presence of toxicities | The presence of toxicies will be monitored through study completion, in an average of 2 years.
  as defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Ow, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Park IH, Ro J, Lee KS, Kim EA, Kwon Y, Nam BH, Jung SY, Lee S, Kim SW, Kang HS. Phase II parallel group study showing comparable efficacy between premenopausal metastatic breast cancer patients treated with letrozole plus goserelin and postmenopausal patients treated with letrozole alone as first-line hormone therapy. J Clin Oncol. 2010 Jun 1;28(16):2705-11. doi: 10.1200/JCO.2009.26.5884. Epub 2010 Apr 26. PMID 20421538
- [Result] Miller TW, Balko JM, Arteaga CL. Phosphatidylinositol 3-kinase and antiestrogen resistance in breast cancer. J Clin Oncol. 2011 Nov 20;29(33):4452-61. doi: 10.1200/JCO.2010.34.4879. Epub 2011 Oct 17. PMID 22010023
- [Result] Massarweh S, Romond E, Black EP, Van Meter E, Shelton B, Kadamyan-Melkumian V, Stevens M, Elledge R. A phase II study of combined fulvestrant and everolimus in patients with metastatic estrogen receptor (ER)-positive breast cancer after aromatase inhibitor (AI) failure. Breast Cancer Res Treat. 2014 Jan;143(2):325-32. doi: 10.1007/s10549-013-2810-9. Epub 2013 Dec 11. PMID 24327334